CLINICAL TRIAL: NCT01073735
Title: Investigating the Needs of Childhood Cancer Survivors: The Unreported Experience
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: INSURE; R21CA142921 (NIH)
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Childhood Cancer
Keywords: Needs assessment; Health-related needs; Childhood cancer survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Survivors: Examine the construct validity, short-term stability, internal consistency and item-response performance of a health-related needs assessment self-report instrument for adult childhood cancer survivors.

SUMMARY:
This feasibility study will determine the psychometric adequacy of a newly developed instrument - Childhood Cancer Survivor Study Needs Assessment Questionnaire (CCSS-NAQ). Additionally, the study will explore the feasibility of selected study methods -- sample selection, length of time to complete recruitment, and response rates - in order to inform a larger national periodic survey of adult survivors' health related needs

DETAILED DESCRIPTION:
This study will focus on the following primary and secondary objectives:

1. Examine the construct validity, short-term stability, internal consistency and item-response performance of a health-related needs assessment self-report instrument for adult childhood cancer survivors
2. Inform future sample stratification by over-sampling minority and rural-dwelling survivors to enhance the heterogeneity of the respondent pool;
3. Describe the met and unmet health-related needs and their covariates in a large, stratified, random sample of childhood cancer survivors;
4. Evaluate the sample selection methods, length of time to complete recruitment, and response rates in the study sample.

ELIGIBILITY:
Inclusion Criteria:

1. Living CCSS participant
2. Age 25 years or older on December 31, 2009
3. History of successful independent (non-surrogate) response to previous CCSS surveys (Flesch-Kincaid reading level for non-medical items established at 4th-6th grade).

Exclusion Criteria:

Received treatment for pediatric malignancy at St. Jude Children's Research Hospital.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be recruited from long-term childhood cancer survivors who are currently participating in the CCSS and whose pediatric malignancy was not treated at St. Jude Children's Research Hospital
Sampling Method: Probability Sample
Enrollment: 1178 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Examine the construct validity, internal consistency, item-response performance, and short-term stability of a health-related needs assessment self-report instrument for adult childhood cancer survivors. | July 2011

SECONDARY OUTCOMES:
Inform future sample stratification by over-sampling minority and rural-dwelling survivors to enhance the heterogeneity of the respondent pool. | July 2011
Describe the met and unmet needs of childhood cancer survivors and their important covariates in a large, stratified random sample of childhood cancer survivors. | July 2011
Evaluate the sample selection methods, length of time to complete recruitment, and response rates in the study sample. | July 2011

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Cox, RN, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org